CLINICAL TRIAL: NCT03953118
Title: A Randomized, Controlled Trial to Evaluate the Role of Oral Azithromycin in the Treatment of Symptomatic Meibomian Gland Disease and Its Effect on the Ocular Surface Microbiome
Brief Title: Azithromycin for Meibomian Gland Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-23877
Record Dates: First submitted 2018-06-27; First posted 2019-05-16 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Dry Eye; Neuropathic Eye Pain; Ocular Microbiome; Depression, Anxiety
MeSH Terms: conditions — Dry Eye Syndromes; Depression; Anxiety Disorders | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Oral
- Azithromycin (Active Comparator)
  Interventions: Drug: Azithromycin Oral Product

INTERVENTIONS:
Drug: Azithromycin Oral Product — Oral azithromycin dosed at 1 gram per week for 3 weeks
  Other Names: Zithromax
  Arms: Azithromycin
Drug: Placebo Oral — Oral placebo tablet
  Arms: Placebo

SUMMARY:
This study aims to elucidate the effectiveness of oral azithromycin in treating symptomatic dry eye syndrome secondary to Meibomian gland dysfunction.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double masked trial of the effectiveness of oral azithromycin in treating symptomatic dry eye syndrome secondary to Meibomian gland dysfunction. Dry eye syndrome (DES) is a persistent feeling of ocular discomfort that encompasses dryness, irritation, foreign body sensation and burning. In the United States, it is the most common non-refractive cause of visits to eye care providers, and has been shown to have a significant impact on quality of life of patients who suffer from this condition. most common cause of DES is Meibomian gland disease (MGD). In the vast majority of cases, MGD is not binding, but rather causes persistant ocular discomfort.

Oral antibiotics, particularly the tetracyclines and macrolides, are frequently prescribed for the treatment of MGD. There is little good-quality evidence to support this practice. This study is designed to evaluate the effectiveness of oral azithromycin on patient-reported dry eye symptoms. Concomitantly, we will also study the composition of the ocular surface microbiome in MGD, and its response for oral antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Meibomian gland disease, defined as patient-reported ocular surface symptoms such as dryness, grittiness, foreign body sensation, or eye fatigue in combination with clinically identifiable Meibomian gland disease with Grade 2 or greater involvement on the Meibomian Gland Grading Scale (Section XV, item 2).
* OSDI Score greater than or equal to 20
* Ability to give informed consent

Exclusion Criteria:

* Age less than 18 years
* Allergy or intolerance to oral azithromycin or topical dexamethasone
* Allergy or intolerance to the preservatives used in topical ophthalmic 0.1% dexamethasone: sodium bisulfite, phenylethyl alcohol, benzalkonium chloride
* History of prolonged QT interval, history of torsades des pointes, congenital long QT syndrome, bradyarrhythmias, heart failure
* Patients currently taking medications that prolong the QT interval (Table 1)
* Aqueous deficiency dry eye defined as Schirmer's strip testing without anesthesia with £ 5mm of tears on two separate tests.
* Ocular surface inflammatory disease, including cicatrizing conjunctivitis, graft versus host disease, Stevens Johnson syndrome
* Atopic disease with ocular involvement
* Limbal stem cell deficiency
* Oral or topical ophthalmic antibiotic use within the last 90 days
* Oral prednisone use >5mg per day
* Topical ophthalmic steroid use within the past 30 days
* Topical ophthalmic anti-inflammatory (including non-steroidal anti-inflammatory medications, lifitegrast, or cyclosporine) use within the past 30 days
* Patients who are currently pregnant, planning on becoming pregnant during the study period, or currently breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Schallhorn, MD, MS, Principal Investigator — University of California, San Francisco; Thuy Doan, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pflugfelder SC. Prevalence, burden, and pharmacoeconomics of dry eye disease. Am J Manag Care. 2008 Apr;14(3 Suppl):S102-6. PMID 18452369
- [Background] The epidemiology of dry eye disease: report of the Epidemiology Subcommittee of the International Dry Eye WorkShop (2007). Ocul Surf. 2007 Apr;5(2):93-107. doi: 10.1016/s1542-0124(12)70082-4. PMID 17508117
- [Background] Schaumberg DA, Nichols JJ, Papas EB, Tong L, Uchino M, Nichols KK. The international workshop on meibomian gland dysfunction: report of the subcommittee on the epidemiology of, and associated risk factors for, MGD. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):1994-2005. doi: 10.1167/iovs.10-6997e. Print 2011 Mar. No abstract available. PMID 21450917
- [Background] Foulks GN, Bron AJ. Meibomian gland dysfunction: a clinical scheme for description, diagnosis, classification, and grading. Ocul Surf. 2003 Jul;1(3):107-26. doi: 10.1016/s1542-0124(12)70139-8. PMID 17075643
- [Background] Knop E, Knop N, Millar T, Obata H, Sullivan DA. The international workshop on meibomian gland dysfunction: report of the subcommittee on anatomy, physiology, and pathophysiology of the meibomian gland. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):1938-78. doi: 10.1167/iovs.10-6997c. Print 2011 Mar. No abstract available. PMID 21450915
- [Background] King-Smith PE, Bailey MD, Braun RJ. Four characteristics and a model of an effective tear film lipid layer (TFLL). Ocul Surf. 2013 Oct;11(4):236-45. doi: 10.1016/j.jtos.2013.05.003. Epub 2013 Jul 12. PMID 24112227
- [Background] Lane SS, DuBiner HB, Epstein RJ, Ernest PH, Greiner JV, Hardten DR, Holland EJ, Lemp MA, McDonald JE 2nd, Silbert DI, Blackie CA, Stevens CA, Bedi R. A new system, the LipiFlow, for the treatment of meibomian gland dysfunction. Cornea. 2012 Apr;31(4):396-404. doi: 10.1097/ICO.0b013e318239aaea. PMID 22222996
- [Background] Lee H, Chung B, Kim KS, Seo KY, Choi BJ, Kim TI. Effects of topical loteprednol etabonate on tear cytokines and clinical outcomes in moderate and severe meibomian gland dysfunction: randomized clinical trial. Am J Ophthalmol. 2014 Dec;158(6):1172-1183.e1. doi: 10.1016/j.ajo.2014.08.015. Epub 2014 Aug 13. PMID 25128594
- [Background] Prabhasawat P, Tesavibul N, Mahawong W. A randomized double-masked study of 0.05% cyclosporine ophthalmic emulsion in the treatment of meibomian gland dysfunction. Cornea. 2012 Dec;31(12):1386-93. doi: 10.1097/ICO.0b013e31823cc098. PMID 23135530
- [Background] Macsai MS. The role of omega-3 dietary supplementation in blepharitis and meibomian gland dysfunction (an AOS thesis). Trans Am Ophthalmol Soc. 2008;106:336-56. PMID 19277245
- [Background] Deinema LA, Vingrys AJ, Wong CY, Jackson DC, Chinnery HR, Downie LE. A Randomized, Double-Masked, Placebo-Controlled Clinical Trial of Two Forms of Omega-3 Supplements for Treating Dry Eye Disease. Ophthalmology. 2017 Jan;124(1):43-52. doi: 10.1016/j.ophtha.2016.09.023. Epub 2016 Nov 3. PMID 27817918
- [Background] Hosseini K, Lindstrom RL, Foulks G, Nichols KK. A randomized, double-masked, parallel-group, comparative study to evaluate the clinical efficacy and safety of 1% azithromycin-0.1% dexamethasone combination compared to 1% azithromycin alone, 0.1% dexamethasone alone, and vehicle in the treatment of subjects with blepharitis. Clin Ophthalmol. 2016 Aug 10;10:1495-503. doi: 10.2147/OPTH.S110739. eCollection 2016. PMID 27570444
- [Background] Greene JB, Jeng BH, Fintelmann RE, Margolis TP. Oral azithromycin for the treatment of meibomitis. JAMA Ophthalmol. 2014 Jan;132(1):121-2. doi: 10.1001/jamaophthalmol.2013.5295. No abstract available. PMID 24201556
- [Background] Yoo SE, Lee DC, Chang MH. The effect of low-dose doxycycline therapy in chronic meibomian gland dysfunction. Korean J Ophthalmol. 2005 Dec;19(4):258-63. doi: 10.3341/kjo.2005.19.4.258. PMID 16491814
- [Background] Ta CN, Shine WE, McCulley JP, Pandya A, Trattler W, Norbury JW. Effects of minocycline on the ocular flora of patients with acne rosacea or seborrheic blepharitis. Cornea. 2003 Aug;22(6):545-8. doi: 10.1097/00003226-200308000-00011. PMID 12883348
- [Background] Wladis EJ, Bradley EA, Bilyk JR, Yen MT, Mawn LA. Oral Antibiotics for Meibomian Gland-Related Ocular Surface Disease: A Report by the American Academy of Ophthalmology. Ophthalmology. 2016 Mar;123(3):492-6. doi: 10.1016/j.ophtha.2015.10.062. Epub 2015 Dec 23. PMID 26707417
- [Background] Watters GA, Turnbull PR, Swift S, Petty A, Craig JP. Ocular surface microbiome in meibomian gland dysfunction. Clin Exp Ophthalmol. 2017 Mar;45(2):105-111. doi: 10.1111/ceo.12810. Epub 2016 Sep 7. PMID 27473509
- [Background] Giamarellos-Bourboulis EJ. Macrolides beyond the conventional antimicrobials: a class of potent immunomodulators. Int J Antimicrob Agents. 2008 Jan;31(1):12-20. doi: 10.1016/j.ijantimicag.2007.08.001. Epub 2007 Nov 1. PMID 17935949
- [Background] Liu Y, Ding J. The combined effect of azithromycin and insulin-like growth factor-1 on cultured human meibomian gland epithelial cells. Invest Ophthalmol Vis Sci. 2014 Aug 14;55(9):5596-601. doi: 10.1167/iovs.14-14782. PMID 25125598
- [Background] Liu Y, Kam WR, Ding J, Sullivan DA. Effect of azithromycin on lipid accumulation in immortalized human meibomian gland epithelial cells. JAMA Ophthalmol. 2014 Feb;132(2):226-8. doi: 10.1001/jamaophthalmol.2013.6030. No abstract available. PMID 24357250
- [Background] Igami TZ, Holzchuh R, Osaki TH, Santo RM, Kara-Jose N, Hida RY. Oral azithromycin for treatment of posterior blepharitis. Cornea. 2011 Oct;30(10):1145-9. doi: 10.1097/ICO.0b013e318207fc42. PMID 21849891
- [Background] Haque RM, Torkildsen GL, Brubaker K, Zink RC, Kowalski RP, Mah FS, Pflugfelder SC. Multicenter open-label study evaluating the efficacy of azithromycin ophthalmic solution 1% on the signs and symptoms of subjects with blepharitis. Cornea. 2010 Aug;29(8):871-7. doi: 10.1097/ICO.0b013e3181ca38a0. PMID 20508503
- [Background] Luchs J. Azithromycin in DuraSite for the treatment of blepharitis. Clin Ophthalmol. 2010 Jul 30;4:681-8. doi: 10.2147/opth.s6370. PMID 20689782
- [Background] Schiffman RM, Christianson MD, Jacobsen G, Hirsch JD, Reis BL. Reliability and validity of the Ocular Surface Disease Index. Arch Ophthalmol. 2000 May;118(5):615-21. doi: 10.1001/archopht.118.5.615. PMID 10815152
- [Background] Korb DR, Blackie CA. Meibomian gland diagnostic expressibility: correlation with dry eye symptoms and gland location. Cornea. 2008 Dec;27(10):1142-7. doi: 10.1097/ICO.0b013e3181814cff. PMID 19034129
- [Background] Meadows JF, Ramamoorthy P, Nichols JJ, Nichols KK. Development of the 4-3-2-1 meibum expressibility scale. Eye Contact Lens. 2012 Mar;38(2):86-92. doi: 10.1097/ICL.0b013e318242b494. PMID 22249431

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Azithromycin
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Study terminated due to lack of funding prior to data collection for for outcomes and adverse events | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Azithromycin | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Ocular Surface Disease Index (OSDI) Questionnaire
Description: Ocular surface disease index - used to evaluate the degree of dry eye symptoms. Scores will range from 0 to 48, where 48 indicates severe dry eye.
Time Frame: Baseline to 1 month
Population: Study terminated prior to data collection for outcomes. No data were collected for this outcome measure.
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Ocular Surface Disease Index (OSDI) Questionnaire
Description: as for outcome 1
Time Frame: Baseline to 3 months
Population: Study terminated prior to data collection for outcomes. No data were collected for this outcome measure.
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Ocular Surface Microbiome Testing
Description: To evaluate the composition of the ocular surface microbiome using Shannon's diversity index. The alpha diversity (local species pool) of the population will be analyzed and compared pre-and post-treatment within and between the azithromycin and control groups. The difference between the bacterial microbiome in the azithromycin and placebo arm will be assessed using a PERMANOVA with an L2 norm distance measure.
  Secondary analyses will include L1 and L0 norms, as well as a phylogenetic distance. In addition, we will assess whether bacterial alpha diversity is decreased in the antibiotic treated arm with the primary outcome being the Simpson's index (L2), with secondary analyses assessing Shannon's (L1) and Richness (L0).
Time Frame: Baseline to 1 month
Population: Study terminated prior to data collection for outcomes. No data were collected for this outcome measure.
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Ocular Surface Microbiome Testing
Description: as for outcome 3
Time Frame: Baseline to 3 months
Population: Study terminated prior to data collection for outcomes. No data were collected for this outcome measure.
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Dry Eye Questionnaire 5 (DE-5)
Description: Dry eye questionnaire 5 - used to evaluate the degree of dry eye symptoms. Scores range from 0-22. A score of 0 represents the minimum dry eye symptoms someone may have and a score of 22 represents the maximum dry eye symptoms someone may have.
Time Frame: Baseline to 1 month
Population: Study terminated prior to data collection for outcomes. No data were collected for this outcome measure.
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Dry Eye Questionnaire 5 (DE-5)
Description: as for outcome 5
Time Frame: Baseline to 3 months
Population: Study terminated prior to data collection for outcomes. No data were collected for this outcome measure.
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Neuropathic Pain Inventory for the Eye (NPSI-E)
Description: Neuropathic pain inventory for the eye - used to study neuropathic vs stimulatory eye pain.
Time Frame: Baseline to 1 month.
Population: study terminated prior to any data analysis
Groups:
- Placebo; Azithromycin: 0
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Neuropathic Pain Inventory for the Eye (NPSI-E)
Description: Neuropathic pain inventory for the eye - used to study neuropathic vs stimulatory eye pain.
Time Frame: Baseline to 3 months
Population: Study terminated prior to data collection for outcomes. No data were collected for this outcome measure.
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Personal Health Questionnaire (PHQ-9)
Description: Personal Health Questionnaire - a brief anxiety and depression questionnaire. Will be used in this study to evaluate the interaction between depression/anxiety and response to treatment.
Time Frame: Baseline to 1 month
Population: Study terminated prior to data collection for outcomes. No data were collected for this outcome measure.
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Personal Health Questionnaire (PHQ-9)
Description: as for outcome 9
Time Frame: Baseline to 3 months
Population: Study terminated prior to data collection for outcomes. No data were collected for this outcome measure.
Arm/Group | Placebo | Azithromycin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected.
Description: Study terminated due to due to lack of funding prior to data collection, adverse events were not monitored.
Arm/Group | Placebo | Azithromycin
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study terminated due to lack of funding prior to data collection for outcome measures and adverse events. There are no data to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-02): https://cdn.clinicaltrials.gov/large-docs/18/NCT03953118/Prot_SAP_000.pdf